CLINICAL TRIAL: NCT00122174
Title: Stress-Busting Program for Caregivers of Patients With Neurological Diseases
Brief Title: Stress-Busting Program for Caregivers of Patients With Neruological Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRI 01-006
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-01

CONDITIONS: Psychological Adaptation; Parkinson's Disease; Neurological Disorders
Keywords: Caregivers; Stress; Coping; Immune; Relaxation; Biofeedback; Bioinstrumentation; Homecare
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Stress Busting Program for family caregivers

INTERVENTIONS:
Behavioral: Stress Busting Program for family caregivers

SUMMARY:
Although family caregivers perform an incredibly valuable service for their relatives and the formal health care system, they do so at a considerable cost to themselves both emotionally and physically. Effective stress management techniques can: 1) help to decrease the caregivers' feelings of burden and stress; 2) improve the emotional and physical health of caregivers; and 3) empower caregivers to gain control of their lives.

DETAILED DESCRIPTION:
The overall goal of this randomized clinical trial is to determine the effectiveness of a stress-busting program (SBP) for caregivers of patients with chronic neurological diseases including stroke, Alzheimer's disease, multiple sclerosis, and Parkinson's disease. Specific research objectives include: 1) Prospectively determine the effects of a SBP compared to a standard support group (SSG) on quality of life and immune response in caregivers of patients with chronic neurological diseases. Subjects will be tested at baseline, at completion of 4 and 8 weeks of SBP or SSG, and at 2- and 4-month follow up sessions. 2) Determine subjects' relaxation response as well as their response to acute laboratory stressors using bioinstrumentation. Muscle tension, electrodermal response, skin temperature, blood volume pulse, and heart rate will be measured. Subjects will be tested at baseline, at completion of 4 and 8 weeks of a SBP or SSG, and at 2- and 4-month follow up sessions. 3) Compare the effectiveness of SBP or SSG for adult children caregivers as compared to spousal caregivers based on quality of life measurements, immune parameters, and relaxation response. The proposed multimodal SBP will focus on a variety of approaches based on cognitive behavioral and relaxation response theories. SBP will consist of a 8-week program with 1�-hour sessions per week. The setting will be an educational support group with topics related to stress, stress and challenges of caregiving, depression, coping strategies, positive thinking, and taking time for oneself. In addition, subjects will be taught simple relaxation strategies that they can practice at home. Outcomes will be measured using psychosocial instruments as well as state-of-the science technology including bioinstrumentation and immune parameters to measure biological responses. Follow up testing will be done 2 and 4 months after the end of the SBP or SSG to determine the long-term effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

The primary caregiver of an individual with a neurological disease. Able to read and converse in English.

Exclusion Criteria:

Presently participating in an ongoing support group related to the neruological disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Questionnaires assessing levels of stress, burden, depression, health, sense of coherence and coping resources; bio-assessment of stress and relaxation, and immune assays. All measures will be taken at baseline, 4 weeks, 8 weeks, 16 weeks, and 32 weeks.

SECONDARY OUTCOMES:
Qualitative data resulting from pre and post intervention interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L. Mantik Lewis, PhD MS BS, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (1):
- South Texas Health Care System, San Antonio, TX, San Antonio, Texas, United States